CLINICAL TRIAL: NCT05681754
Title: Endodontic-periodontal Disease - Comparison of Treatment Outcome Using Conventional and Hydraulic Calcium Silicate Sealer With or Without LPRF and Characterisation of Host-microbiome Interaction
Brief Title: Endo-perio Disease - Treatment Outcomes Using Conventional and Hydraulic Calcium Silicate Sealer With or Without LPRF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDGE 147667
Record Dates: First submitted 2022-12-16; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Endodontic Disease; Periodontitis
Keywords: Endo-perio lesions
MeSH Terms: conditions — Dental Pulp Diseases; Periodontitis | interventions — Bone Substitutes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Operators for endodontic - periodontal treatment will be different from the assessors for the initial assessments and subsequent review appointments.
  The Treatment will be masked for the patient and assessor. As the blood samples will be collected from the patients at T6 for biomarker analysis, therefore the patient can be masked about the treatment as these blood can be used for the LPRF treatment for those patient who are randomised in the LPRF group.
  The statistician will also be blinded to the allocations and will only conduct the analysis in a semi-blinded way (group 1 vs group 2 vs group 3 vs group 4) without knowing the corresponding groups until the analysis is complete.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RCT using hydraulic calcium silicate sealer and L-PRF + GTR (Experimental): Endodontic-periodontal disease patients undergoing root canal treatment using hydraulic calcium silicate sealer and L-PRF + GTR (bone substitute + collagen membrane)
  Interventions: Procedure: Experimental: RCT using hydraulic calcium silicate sealer and L-PRF + GTR
- RCT using conventional sealer and L-PRF + GTR (Experimental): Endodontic-periodontal disease patients undergoing root canal treatment using conventional sealer and L-PRF + GTR (bone substitute + collagen membrane)
  Interventions: Procedure: Experimental: RCT using conventional sealer and L-PRF + GTR
- RCT using hydraulic calcium silicate sealer and GTR (Experimental): Endodontic-periodontal disease patients undergoing root canal treatment using hydraulic calcium silicate sealer and GTR (bone substitute + collagen membrane)
  Interventions: Procedure: Experimental: RCT using hydraulic calcium silicate sealer and GTR
- RCT using conventional sealer and GTR (bone substitute + collagen membrane) (Active Comparator): Endodontic-periodontal disease patients undergoing root canal treatment using conventional sealer and GTR (bone substitute + collagen membrane)
  This is our control group Both the endodontic and periodontal lesions are managed using gold standard of care biomaterials and techniques
  Interventions: Procedure: Active Comparator: RCT using conventional sealer and GTR (bone substitute + collagen membrane)

INTERVENTIONS:
Procedure: Experimental: RCT using hydraulic calcium silicate sealer and L-PRF + GTR — Endodontic treatment with hydraulic calcium silicate sealer, followed by periodontal surgery using GTR +/- LPRF
  Arms: RCT using hydraulic calcium silicate sealer and L-PRF + GTR
Procedure: Experimental: RCT using conventional sealer and L-PRF + GTR — Endodontic treatment with conventional sealer followed by periodontal treatment with PRF + GTR
  Arms: RCT using conventional sealer and L-PRF + GTR
Procedure: Experimental: RCT using hydraulic calcium silicate sealer and GTR — Endodontic treatment with hydraulic calcium silicate sealer, followed by periodontal surgery using GTR only
  Arms: RCT using hydraulic calcium silicate sealer and GTR
Procedure: Active Comparator: RCT using conventional sealer and GTR (bone substitute + collagen membrane) — Endodontic treatment with conventional sealer followed by periodontal treatment with GTR only
  Arms: RCT using conventional sealer and GTR (bone substitute + collagen membrane)

SUMMARY:
The endodontic periodontal-disease is characterized by the involvement of the pulp and periodontal disease in the same tooth. The anatomic connections between the dental pulp and the periodontium provide a pathway for perio-endo communication via apical foramina, lateral canals, exposed dentinal tubules, and developmental grooves. These pathways provide an egress for pulpal disease to affect the periodontium and conversely, an ingress for periodontal disease to affect the pulp.

Teeth with endo-perio disease, which are deemed salvageable might require root canal (endodontic) treatment, followed by staged periodontal treatment. Compared to conventional sealers used for endodontic treatment, the hydraulic calcium silicate based sealers (HCSB)s have excellent sealing ability, biocompatibility, regeneration ability, and antimicrobial characteristics. However little is known about its clinical benefits when used to treat endo-perio disease.

The gold standard treatment for periodontitis affected teeth associated with intrabony lesions is guided tissue regeneration (GTR) which has significant improved clinical outcomes over open flap debridement (Cochrane systematic review 2005). However, the success the of this regenerative technique requires careful case and defect selection. We propose the use of an autologous bioactive scaffold, leukocyte platelet rich fibrin (L-PRF) to achieve regeneration of periodontal soft and hard tissues, resulting in faster healing, greater bone infill and improved predictability of clinical outcomes

DETAILED DESCRIPTION:
Primary periodontal /secondary endodontic lesions and true combined lesions is challenging since the outcome of these is significantly less predictable than that of those arising due to primary endo disease and require multidisciplinary management involving endodontic treatment in the form of root canal treatment followed by staged periodontal treatment.

This includes initial non-surgical periodontal therapy to reduce the microbiologic burden in the periodontal pocket. After a 3-to-6 month period following the completion of endodontic treatment, the apical healing is evaluated and the periodontal condition reassessed and then the decision is made for periodontal regenerative therapies to promote the formation of new cementum, periodontal ligament, and bone to achieve esthetic and hygienic goals. These regenerative therapies include tissue engineering techniques, such as guided tissue regeneration (GTR); implantation of enamel protein matrix derivatives; application of signalling molecules, such as growth factors, and leucocyte- platelet rich fibrin (L-PRF). Without concomitant regenerative procedures, success ranges from 27% to 37%. When regenerative procedures are added to endodontic therapy, the chance of a successful outcome improves to 77.5%.

L-PRF is obtained through the centrifugation of blood resulting in a strong fibrin matrix enriched with platelets and growth factors. Previous evidence suggest that this can be successfully used in the treatment of intrabony defects, but no randomised controlled trial has been conducted examining the additional benefits of L-PRF when used in conjunction with GTR in the treatment of intrabony defects associated with endodontic-periodontal disease.

The investigators have previously also investigated the microbiome of endodontic infections using targeted 16SrRNA gene and house-keeping gene sequence analysis, we determined the predominant cultivable microbiota of primary and secondary (failed) Endodontic infections. The investigators have lately investigated the microbiome of root canal infections using next generation sequencing targeting region V1-V2 of 16SrRNA gene (unpublished data). The investigators are also currently investigating the host microbiome interactions in these conditions. Although Endodontic periodontal disease differ in pathogenicity but they do share common microbial factors and inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of Endodontic-periodontal disease without root damage in periodontitis patients, Grades I, II, III according to Herrera 2017 classification.

  * Presence of ≥ 1 intrabony defect: interproximal probing pocket depth ≥ 5 mm and ≥ 3mm radiographic intrabony defect, adjacent to single rooted and multi-rooted teeth associated with endodontic-periodontal disease
  * Age: 18-80
  * Non-smokers (zero cigarettes within last 5 years)

Exclusion Criteria:

* Endodontic considerations: severely sclerosed canals, external cervical resorption and internal root resorption, perforations, root fracture or cracking, re- RCT, apical surgery and unrestorable teeth
* Teeth with defects not amenable to regeneration or molar teeth planned for root resection

  - Periodontal treatment carried out previously to the study site within the last 12 months (excluding not-extensive subgingival debridement as judged by the examining clinician),
* presence of drug induced gingival overgrowth.
* Smoking (current or in past 5 years) including e-cigarettes/ vaping
* History of alcohol or drug abuse,
* Systemic antibiotic therapy during the 3 months preceding the baseline exam,
* History of conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures,
* Anti-inflammatory or anticoagulant therapy during the month preceding the baseline exam,
* Medical history of diabetes or transmittable diseases,
* Chronic inflammatory conditions: chronic peptic ulcer, tuberculosis, rheumatoid arthritis, ulcerative colitis, crohn's disease, active hepatitis, inflammatory bowel diseases, irritable bowel syndrome, autoimmune diseases, liver diseases, renal diseases or cancer
* Medications which alter bone metabolism: hormone replacement therapy, immunosuppressive drugs, corticosteroids, selective serotonin reuptake inhibitors, tumour necrosis factor blockers, IV bisphosphonates, and/or antiresorptive drugs,
* Self-reported pregnancy or lactation
* Surgical procedures in the last 6months (any type of surgical procedures)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that according to the investigator may increase the risk associated with trial participation,
* Poor compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth change in mm | at 12months (T8); at 18months (T9)
  Probing pocket depth change in mm at 12months (T8); at 18months (T9)
Clinical attachment level (CAL) change in mm | at 12months (T8); at 18months (T9)
  Clinical attachment level (CAL) change in mm at 12months (T8); at 18months (T9)
Change in the size of the lesion/ intrabony defect using Cone Beam CT and PA radiographs. | at 12months (T8); at 18months (T9)
  Change in the size of the lesion/ intrabony defect using Cone Beam CT and PA at 12months (T8); at 18months (T9)

SECONDARY OUTCOMES:
Changes in levels of inflammatory markers and growth factors in blood, saliva and GCF (T1, T2, T3, T5, T7, T8, T9) | baseline (T1), Endodontic treatment, within 4 weeks from baseline (T2), Review at 3months (T3), Review at 6 months (T5), Review at 9 months (T7), Review at 12months( T8), Review at 18months (T9)
  Changes in levels of inflammatory markers and growth factors in blood, saliva and GCF (T1, T2, T3, T5, T7, T8, T9)
Plaque, Salivary and root canal microbiome associated with presence and healing of intrabony defects (T1, T2, T3, T5, T7, T8, T9) | baseline (T1), Endodontic treatment, within 4 weeks from baseline (T2), Review at 3months (T3), Review at 6 months (T5), Review at 9 months (T7), Review at 12months( T8), Review at 18months (T9)
  Plaque, Salivary and root canal samples for microbiome analysis
Expression of inflammatory mediators from granulation tissue derived from periodontal intrabony defects (T6) | Surgical periodontal treatment, within 6-8 months from endodontic treatment (T6)
  Expression of inflammatory mediators from granulation tissue derived from periodontal intrabony defects (T6)
Patient reported outcome measures (PROMs) | baseline (T1), Endodonic treatment, within 4 weeks from baseline (T2), Review at 3months (T3), Review at 6 months (T5), Review at 9 months (T7), Review at 12months( T8), Review at 18months (T9)
  This will be measured using standardised questionnaire, the Oral Health Impact Profile short form (OHIP-14)

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Niazi, Principal Investigator — King's College London, London SE1 9RT
Locations (1):
- Guy'S and St Thomas' Nhs Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The research data will only be accessed by PIs, or CIs involved in the research project. The PhD student and statistician will only have access to anonymised data